CLINICAL TRIAL: NCT03088774
Title: Comparing Satisfaction With a Participatory Driven Web-application and a Standard Website for Patients With Low Back Pain: a Study Protocol of a Randomised Controlled Trial
Brief Title: Comparing Satisfaction With a Participatory Driven Web-application and a Standard Website
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary trial was stopped. Since, a feasibility study showed that recruitment was not feasible. We obtain a recruitment rate of 15 %.
Sponsor: Aalborg University Hospital (Other)
Collaborators: The Novo Nordic Foundation (Other); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Allan Riis, Post doc, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AllanRiis_4
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Allocation of patients 1:1 to the new web-application or to Patient's Handbook
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation sequence will be delivered by the statistician group at Aalborg University Hospital and delivered to a IT consultant at ProData (Viby, J, Denmark) and integrated in the web-application. The researchers conducting the analysis will be blinded. During the project, data will be stored on a server placed at Aalborg University. Another member of the author Group will prepare a data set with a dummy variable for allocation without free text information from patients and make this data set available for the assessors to analyse. Patients will be aware of their allocation. General practitioners will only be aware of the allocation if the patient chooses to tell it to the general practitioner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New web-application (Experimental): Information material developed in a participatory design together with patients.
  Interventions: Other: Information material
- Patient Handbook (Experimental): Public available information.
  Interventions: Other: Information material

INTERVENTIONS:
Other: Information material — Online web-application developed together with patients with low back pain

SUMMARY:
This project studies the effects of involving patients in the development of a web-application.

DETAILED DESCRIPTION:
The point-prevalence of low back pain (LBP) has been estimated to 9.4 % and LBP is in many countries the most frequent reason to consult a general practitioner. However, general practitioners are under pressure with increasing workloads. The increasing number of patients and the typical 10-15 minutes of available time for each patient are challenging the provision of sufficient information and advice. According to international guidelines information and advice are recommended for every patient with LBP, therefore, new methods to support general practitioners (GPs) are very much needed. Online technologies give new opportunities to extend the treatment. Furthermore, involving patients with LBP in the development of online information material may produce more user friendly content and design and thereby increasing patients' acceptance and usage. Thus, optimizing clinical outcome. This project will study patients' satisfaction and clinical outcomes of a web-application for patients with LBP consulted in general practice compared to best existing technology (the Patient Handbook).

ELIGIBILITY:
Inclusion Criteria:

* Contacting general practice with low back pain

Exclusion Criteria:

* Spinal stenosis
* Spine fractures
* Cauda equina syndrome
* Spinal malignancy
* Osteoporosis
* Spondyloarthritis
* Without Danish reading skills
* Without internet access
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
General satisfaction | 12 weeks
  The question: 'how likely is it that you would recommend this web-application to a friend or colleague?' will be applied to measure satisfaction. The patients will be asked to choose between 11 boxes displayed on a horizontal line (10-0 Points, higher score indicating more satisfaction). The scales will be labelled to the left at 10 (extremely likely) and at the right side as 0 (not at all likely). It is only possible to tick off one box, if the patient change decision while filling in the online questionnaire, another box can be ticked off and the first choice will automatically delete. Responses of 10-9 are grouped as 'satisfied' of the web-application and patients replying 8-0 will be grouped as 'not satisfied'. The proportion of patients being satisfied after 12 weeks is the primary analysis. The proportion of patients being satisfied after 1, 2, 4, and 8 weeks will be carried out as secondary analyses.

SECONDARY OUTCOMES:
Functional improvement | 12 weeks
  Roland Morris functional disability score (RMDQ, the Patrick version, 0-23 points)
Pain intensity | 1, 2, 4, 8, and 12 weeks
  Numerical pain rating of current pain (0-10 Points, rating from 'no pain' to 'maximal pain' )
Improvement in self-rated health | 12 weeks
  EQ-5D-5L (EuroQol - 5 Diminsions - 5 Levels)
Employment status | 12 weeks
  Self reported current employment status (yes/no)
Sick leave | 12 weeks
  Self reported number of hours of sick leave during the study
Contacts to general practice | 12 weeks
  Self reported number of general practice contacts since study inclusion
Contacts to primary care physiotherapists | 12 weeks
  Self reported number of physiotherapy contacts since study inclusion
Contacts to primary care chiropractors | 12 weeks
  Self reported number of chiropractor contacts since study inclusion
Contacts to secondary care | 12 weeks
  Contact to secondary care because of low back pain during the study (yes/no)
Cost utility analysis | 12 weeks
  A analysis comparing the intervention group with the control group from a healthcare perspective. Including primary care costs such as public paid costs for GP contacts, physiotherapy services, and chiropractic services. Quality adjusted life years (QALYs) will be applied as measure of effect based on EQ-5D-5L. We will not include costs for developing and maintaining the new technology or other protocol driven costs. Based on the relative short time-horizon costs and effects will not be discounted.
Specific satisfaction | 1, 2, 4, 8, and 12 weeks
  For further exploration of reasons for the primary outcome we include a question regarding the general satisfaction with the web-application (10-0) and detailed questions/items regarding satisfaction with design (very, some, little, none), satisfaction with customisation (very, some, little, none ), satisfaction with usability (very, some, little, none ), satisfaction with readability (very, some, little, none), and satisfaction with credibility (very, some, little, none). It is only possible to tick off one box to each item, if the patient change decision while filling in the online questionnaire, another box can be ticked off and the first choice will automatically delete. Furthermore, these items will be validated against the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Riis, PhD, Principal Investigator — Research unit for General Practice in Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riis A, Rathleff MS, Hartvigsen J, Thomsen JL, Afzali T, Jensen MB. Feasibility study on recruitment in general practice for a low back pain online information study (part of the ADVIN Back Trial). BMC Res Notes. 2020 Jan 10;13(1):24. doi: 10.1186/s13104-020-4894-8. PMID 31924258
- [Derived] Riis A, Hartvigsen J, Rathleff MS, Afzali T, Jensen MB. Comparing satisfaction with a participatory driven web-application and a standard website for patients with low back pain: a study protocol for a randomised controlled trial (part of the ADVIN Back Trial). Trials. 2018 Jul 25;19(1):399. doi: 10.1186/s13063-018-2795-0. PMID 30045749